CLINICAL TRIAL: NCT01537562
Title: Early Versus Delayed Insertion of Intrauterine Contraception After Medical Abortion- a Randomized Controlled Trial
Brief Title: Intrauterine Contraception (IUC) After Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, Professor, Head of Department, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WIUC12
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: IUC Insertion After Medical Abortion
Keywords: Copper IUD; LNG-IUS; intrauterine contraception; medical abortion; postabortion contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delayed IUC insertion (Active Comparator): Patients randomised to delayed, routine, insertion had their IUC inserted at 3-4 weeks (day 21-35 after mifepristone treatment
  Interventions: Other: Timing of IUC insertion
- Early IUC insertion (Active Comparator): Patients randomised to early insertion had their IUC inserted on day 5-9 after mifepristone treatment.
  Interventions: Other: Timing of IUC insertion

INTERVENTIONS:
Other: Timing of IUC insertion — Patients randomised to early insertion had their IUC inserted on day 5-9 after mifepristone treatment while patients randomised to delayed insertion had the IUC insertion at about 3 to 4 weeks after mifepristone.
  Other Names: Women were free to chose the type of IUC

SUMMARY:
Today a large proportion of early abortions are medical, in accordance to the woman's choice. The main objective of the present study was to compare, in a randomised fashion, initiation of intrauterine contraception (IUC) at about 1 week versus 3 to 4 weeks post medical abortion with regard to expulsions and safety.

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* elective medical abortion up to 9 weeks (63 days) of amenorrhea
* general good health and
* good understanding of Swedish language.

Exclusion Criteria:

* pathological pregnancies or abnormality of the uterus
* complications after the medical abortion, such as on-going pregnancy retained gestational sac or endometritis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2007-02; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Expulsion | 6 months after IUC insertion
  Expulsions are recorded up to 6 months after the IUC insertion

SECONDARY OUTCOMES:
PID | within 6 months of IUC insertion
  Pelvic inflammatory disease reported or diagnosed at FU
serum hemoglobin | 4 weeks post IUC insertion
  S-Hb was measured at IUC insertion and at 4 weeks post insertion
Compliance | 6 months
  impact on the number of women who return for IUC insertion, and compliance with IUC use during the first 6 months following insertion
Bleeding patterns | 4 weeks
  Bleeding patterns during the first 4 weeks post IUC insertion

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, MD, PhD, Principal Investigator — WHO centre, Dept of Women's and Childrens' Health, Div of Obstetrics and Gynecology, Karolinska Institutet/ Karolinska Univeristy Hospital
Locations (1):
- WHO centre, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Saav I, Stephansson O, Gemzell-Danielsson K. Early versus delayed insertion of intrauterine contraception after medical abortion - a randomized controlled trial. PLoS One. 2012;7(11):e48948. doi: 10.1371/journal.pone.0048948. Epub 2012 Nov 14. PMID 23155432